CLINICAL TRIAL: NCT01795482
Title: The Effect of Preoperative Patient Warming in the Prevention of Perioperative Hypothermia in Major Abdominal Surgery Under Combined General/Epidural Anaesthesia
Brief Title: Preoperative Patient Warming for Prevention of Perioperative Hypothermia in Major Abdominal Surgery
Acronym: THER-6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, PD Dr. Jan Hoecker, Associate Professor of Anaesthesiology, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THER-6
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Preoperative Warming; Prewarming; Perioperative Hypothermia; General Anaesthesia; Epidural Anaesthesia; Temperature Monitoring
Keywords: perioperative hypothermia; prewarming; preoperative warming; general anaesthesia; epidural anaesthesia; temperature measurement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 2, Prewarming only before general anaesthesia (Experimental): Active forced-air warming for 15 min after completion of epidural anaesthesia / before start of general anaesthesia. Continued active forced-air warming after induction of general anaesthesia until operation is finished (intraoperatively). Application of warmed infusions (41 °C).
  Interventions: Device: Forced-air warming
- Group 3, Prewarming before epidural and general anaesthesia (Experimental): Active forced-air warming for 15 min before start of epidural anaesthesia and for 15 min after completion of epidural anaesthesia / before start of general anaesthesia. Continued active forced-air warming after induction of general anaesthesia until operation is finished (intraoperatively). Application of warmed infusions (41 °C).
  Interventions: Device: Forced-air warming
- Group 1, control group (No Intervention): No active warming before start of epidural or general anaesthesia, active forced-air warming after induction of general anaesthesia until operation is finished (intraoperatively). Application of warmed infusions (41 °C).

INTERVENTIONS:
Device: Forced-air warming — In the intervention groups a forced-air cover (Level 1 Snuggle Warm Upper Body Blanket, Smiths Medicals) will be positioned over the patients sitting or laying on the operating table for 15 min before start of epidural anaesthesia and afterwards till start of general anaesthesia (group 3), for 15 min before start of general anaesthesia (group 2) or only after induction of general anaesthesia (group 1, control). All patients will receive forced-air warming after induction of general anaesthesia till end of surgery.
  Other Names: Level 1 Snuggle Warm Upper Body Blanket; Forced-air warming blower
  Arms: Group 2, Prewarming only before general anaesthesia; Group 3, Prewarming before epidural and general anaesthesia

SUMMARY:
The study should evaluate how long patients undergoing major abdominal surgery under combined general/epidural anaesthesia have to be actively warmed preoperatively to prevent perioperative hypothermia and postoperative shivering. 99 patients will receive forced-air skin-surface warming for different duration. Body temperature will be measured at the tympanic membrane. The investigators hypothesize that active warming before starting the epidural anaesthesia will decrease the incidence of perioperative hypothermia.

DETAILED DESCRIPTION:
The aim of our study is to evaluate the performance of different durations of active preoperative skin-surface warming (prewarming) to prevent perioperative hypothermia in patients undergoing major abdominal surgery under combined general/epidural anaesthesia. The investigators plan to enroll 99 patients in 3 groups. Body temperature will be measured at the tympanic membrane. The investigators hypothesize that active warming before starting the epidural anaesthesia will decrease the incidence of perioperative hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* planned duration of surgery > 2 hours
* planned for elective major abdominal surgery under combined epidural/general anaesthesia
* written informed consent
* American society of anesthesiologists status 1-3

Exclusion Criteria:

* duration of surgery < 90 min
* withdrawal of consent
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of hypothermic patients at arrival at PACU | 2 hours
  After the operation patients will be admitted to the PACU. Here, body temperature will be assessed and the incidence of hypothermic patients (body temperature < 36°C)will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hoecker, M.D., Study Chair — University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany
Locations (2):
- Germany (2):
  - University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - Klinikum Pinneberg Klinik für Anästhesiologie, Intensivmedizin und OP-Management, Pinneberg, Schleswig-Holstein

REFERENCES:
- [Background] Horn EP, Bein B, Bohm R, Steinfath M, Sahili N, Hocker J. The effect of short time periods of pre-operative warming in the prevention of peri-operative hypothermia. Anaesthesia. 2012 Jun;67(6):612-7. doi: 10.1111/j.1365-2044.2012.07073.x. Epub 2012 Feb 29. PMID 22376088
- [Background] Hocker J, Bein B, Bohm R, Steinfath M, Scholz J, Horn EP. Correlation, accuracy, precision and practicability of perioperative measurement of sublingual temperature in comparison with tympanic membrane temperature in awake and anaesthetised patients. Eur J Anaesthesiol. 2012 Feb;29(2):70-4. doi: 10.1097/EJA.0b013e32834cd6de. PMID 22037543
- [Derived] Horn EP, Bein B, Broch O, Iden T, Bohm R, Latz SK, Hocker J. Warming before and after epidural block before general anaesthesia for major abdominal surgery prevents perioperative hypothermia: A randomised controlled trial. Eur J Anaesthesiol. 2016 May;33(5):334-40. doi: 10.1097/EJA.0000000000000369. PMID 26555870